CLINICAL TRIAL: NCT03650400
Title: A Multicenter, Open-label, 8 Day Treatment Study to Assess the Pharmacokinetics, Safety and Tolerability of Fevipiprant Delivered Via a Once Daily Chewable Tablet in Children Aged 6 to <12 Years With Asthma
Brief Title: Pharmacokinetics, Safety and Tolerability of Fevipiprant Delivered Via a Once Daily Chewable Tablet in Children Aged 6 to < 12 Years With Asthma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company Decision
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CQAW039B2201
Record Dates: First submitted 2018-08-27; First posted 2018-08-28 (Actual); Results first posted 2020-07-20 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Asthma
Keywords: Fevipiprant,; GINA 2018,; Pediatrics
MeSH Terms: conditions — Asthma | interventions — fevipiprant

STUDY DESIGN:
Intervention Model Description: There will be 2 treatment dose cohorts studied (fevipiprant dose A once daily and one higher dose selected based on PK obtained at dose A mg/day, fevipiprant dose B once daily). Within each dose cohort, subjects will be stratified approximately 1:1 ratio into 2 age groups: ages 6 to < 9 years and ages 9 to < 12 years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort A Fevipiprant 75 mg (Experimental): QAW039 75 mg Chewable tablet
  Interventions: Drug: Fevipiprant
- Cohort B Feviprant 375 mg (Experimental): QAW039 375 mg Chewable tablet
  Interventions: Drug: Fevipiprant

INTERVENTIONS:
Drug: Fevipiprant — Chewable tablet
  Other Names: QAW039

SUMMARY:
The purpose of this study was to assess the pharmacokinetics (PK) of fevipiprant (QAW039) delivered as a chewable tablet (CT) in pediatric asthma subjects aged 6 to < 12 years with asthma. The results of this study will support the identification of a fevipiprant dose for subsequent pediatric efficacy studies aiming to provide an exposure similar to that of the to-be marketed adult/adolescent dose. In addition, the first data on safety and tolerability of fevipiprant in this age group was obtained.

DETAILED DESCRIPTION:
The purpose of this study was to assess the pharmacokinetics (PK) of fevipiprant delivered as a chewable tablet (CT) in pediatric asthma subjects aged 6 to < 12 years. The results of this study would have supported the identification of a fevipiprant dose for subsequent pediatric efficacy studies aiming to provide an exposure similar to that of the to-be marketed adult/adolescent dose. Based on evaluation of the fevipiprant asthma development program in the recently completed studies (CQAW039A2307/ CQAW039A2314) in the adult population (the analyses of these studies did not meet the clinically relevant threshold for reduction in rate of moderate-to-severe exacerbation compared to placebo over a 52-week treatment period for either of the doses [i.e. 150 mg/ 450 mg]), Novartis decided to discontinue this study (CQAW039B2201).

ELIGIBILITY:
Inclusion Criteria:

* Children
* Written informed consent by parent(s)/legal guardian(s) for the pediatric patient and assent by the pediatric patient (depending on local requirements) must be obtained before any study-specific assessment is performed.
* Confirmed/documented diagnosis of asthma, as defined by national or international asthma guidelines for at least 6 months prior to study enrollment.
* Subjects using asthma rescue medication (e.g. SABA) without asthma controller therapy or patients receiving daily treatment with a stable dose ICS (with or without additional controller such as long-acting β-agonists (LABA), long-acting muscarinic antagonists (LAMA)) for at least 4 weeks prior to Treatment Visit (Day 1).
* Subjects must be able to attend study visits as per Study Visit Assessment Schedule (Section 8) which includes 8 to 9 hours in the clinic/home on the day of End of Treatment Visit and have blood draws as scheduled in the study.

Exclusion Criteria:

* Use of other investigational drugs within 5 half-lives of enrollment, or (within 30 days (for small molecules)/until the expected pharmacodynamic effect has returned to baseline (for biologics)), whichever is longer.
* Subject is unable to ingest banana and/or yogurt
* History of hypersensitivity to any of the study drugs or its excipients or to drugs of similar chemical classes.
* History of chronic lung disease other than asthma such as and not limited to, sarcoidosis interstitial lung disease, cystic fibrosis, mycobacterial or other infection (including active tuberculosis or atypical mycobacterial disease).
* History of active bacterial, viral or fungal infection within 6 weeks of Treatment Visit (Day 1).

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2019-12-16 (Actual); Study Completion 2020-01-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- United States (6):
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, Columbia, Missouri
  - Novartis Investigative Site, Tulsa, Oklahoma
  - Novartis Investigative Site, Boerne, Texas
  - Novartis Investigative Site, El Paso, Texas
  - Novartis Investigative Site, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com https://www.clinicalstudydatarequest.com/
URL: https://www.clinicalstudydatarequest.com/

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=846
- See also: A Pediatric Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=486

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Six US centers recruited 11 subjects in the study.
Pre-assignment Details: A total of 19 subjects were screened to enroll 11 subjects in the study
Period: Overall Study
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg
Started | 6 | 5
Completed | 6 | 0
Not Completed | 0 | 5
Not completed — Study terminated by sponsor | 0 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (1.83) | 9.4 (1.52) | 8.7 (1.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 4 | 10
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics of Fevipiprant by Area Under the Curve From 0 to 24 Hours at Steady State (AUC0-24h,ss), After at Least Four Consecutive Days of Dosing
Description: Area under the curve (AUC0-24h,ss), steady state following drug administration
Time Frame: End of Treatment (pre-dose, 0.5hours, 1 hour, 2 hours, 3 hours, 5 hours and 8 hours)
Population: All treated participants with a valid PK measurement. No PK samples were collected for PK analysis in Cohort B due to early study termination.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg
Number analyzed (Participants) | 6 | 0
h*ng/mL | 2380 (1880) |

2. Primary Outcome: Pharmacokinetics of Fevipiprant by Maximum Plasma Concentration at Steady State (Cmax,ss), After at Least Four Consecutive Days of Dosing
Description: Maximum plasma concentration (Cmax,ss) steady state following drug administration.
Time Frame: End of Treatment (pre-dose, 0.5hours, 1 hour, 2 hours, 3 hours, 5 hours and 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg
Number analyzed (Participants) | 6 | 0
ng/mL | 394 (286) |

3. Primary Outcome: Pharmacokinetics of Fevipiprant by Oral Clearance at Steady State (CL/F), After at Least Four Consecutive Days of Dosing
Description: Oral clearance (CL/F), steady state following drug administration.
Time Frame: End of Treatment (pre-dose, 0.5hours, 1 hour, 2 hours, 3 hours, 5 hours and 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg
Number analyzed (Participants) | 6 | 0
L/h | 48.2 (32) |

4. Secondary Outcome: Pharmacokinetics of Fevipiprant by CL/F
Description: Pharmacokinetics of fevipiprant by oral clearance (CL/F) at steady state
Time Frame: End of Treatment (pre-dose, 0.5hours, 1 hour, 2 hours, 3 hours, 5 hours and 8 hours.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg
Number analyzed (Participants) | 6 | 0
L/h | 48.2 (32.0) |

5. Secondary Outcome: Pharmacokinetics of Fevipiprant by Tmax,ss
Description: Pharmacokinetics of fevipiprant by time of maximum plasma concentration (Tmax,ss) at steady state
Time Frame: End of Treatment (pre-dose, 0.5hours, 1 hour, 2 hours, 3 hours, 5 hours and 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg
Number analyzed (Participants) | 6 | 0
h | 1.42 (0.916) |

6. Secondary Outcome: Urinary Excretion of Fevipiprant
Description: CLr, amount and fraction of dose excreted over the PK collection interval at steady state, of fevipiprant
Time Frame: End of Treatment (pre-dose, 0.5hours, 1 hour, 2 hours, 3 hours, 5 hours and 8 hours.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg
Number analyzed (Participants) | 6 | 0
L/h | 6.61 (4.88) |

7. Secondary Outcome: Pharmacokinetics of Fevipiprant by Cmin,ss
Description: Pharmacokinetics of fevipiprant by minimum plasma concentration (Cmin,ss) at steady state
Time Frame: End of Treatment (pre-dose, 0.5hours, 1 hour, 2 hours, 3 hours, 5 hours and 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg
Number analyzed (Participants) | 6 | 0
ng/mL | 28.3 (13.8) |

8. Secondary Outcome: Pharmacokinetics of the Metabolite CCN362 by AUC0-24h,ss
Description: Pharmacokinetics of CCN362 metabolite of fevipiprant , area under the curve (AUC0-24h,ss) at steady state.
Time Frame: End of Treatment (pre-dose, 0.5hours, 1 hour, 2 hours, 3 hours, 5 hours and 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg
Number analyzed (Participants) | 6 | 0
h*ng/mL | 2760 (1210) |

9. Secondary Outcome: Pharmacokinetics of the Metabolite CCN362 by Cmax,ss
Description: Pharmacokinetics of CCN362 metabolite of fevipiprant by maximum plasma concentration (Cmax,ss) at steady state
Time Frame: End of Treatment (pre-dose, 0.5hours, 1 hour, 2 hours, 3 hours, 5 hours and 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg
Number analyzed (Participants) | 6 | 0
ng/mL | 302 (134) |

10. Secondary Outcome: Pharmacokinetics of the Metabolite CCN362 by Cmin,ss
Description: Pharmacokinetics of CCN362 metabolite of fevipiprant by minimum plasma concentration (Cmin,ss) at steady state
Time Frame: End of Treatment (pre-dose, 0.5hours, 1 hour, 2 hours, 3 hours, 5 hours and 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg
Number analyzed (Participants) | 6 | 0
ng/mL | 33.6 (22.6) |

11. Secondary Outcome: Pharmacokinetics of the Metabolite CCN362 by Tmax,ss
Description: Pharmacokinetics of CCN362 metabolite of fevipiprant by time of maximum plasma concentration (Tmax,ss) at steady state
Time Frame: End of Treatment (pre-dose, 0.5hours, 1 hour, 2 hours, 3 hours, 5 hours and 8 hours)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg
Number analyzed (Participants) | 6 | 0
h | 2.69 (1.20) |

12. Secondary Outcome: Urinary Excretion of the Metabolite, CCN362
Description: CLr, amount and fraction of dose excreted over the PK collection interval at steady state, of the metabolite, CCN362
Time Frame: End of Treatment (pre-dose, 0.5hours, 1 hour, 2 hours, 3 hours, 5 hours and 8 hours.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg
Number analyzed (Participants) | 6 | 0
L/h | 5.10 (1.96) |

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) are presented from first dose of study treatment until last dose of study treatment plus 7 days post treatment. Serious AEs are presented from first dose of study treatment until last dose of study treatment plus 30 days post treatment, up to maximum duration of 38 weeks.
Arm/Group | Cohort A Fevipiprant 75 mg | Cohort B Feviprant 375 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2019-02-13): https://cdn.clinicaltrials.gov/large-docs/00/NCT03650400/Prot_001.pdf
  • Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT03650400/SAP_000.pdf